CLINICAL TRIAL: NCT01028560
Title: Efficacy of Allergy Immunotherapy in Preventing Asthma Morbidity in Atopic, Wheezing Children (Age 18 Months - 3 Years)
Brief Title: Allergy Immunotherapy for the Reduction of Asthma
Acronym: AIR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Jacobi Medical Center (Other)
Responsible Party: Principal Investigator, Gabriele de Vos, Assistant Professor of Medicine (Allergy and Immunology), Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-280
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-04

CONDITIONS: Wheezing; Asthma; Allergy
Keywords: Wheezing; Asthma; Allergy; Immunotherapy
MeSH Terms: conditions — Respiratory Sounds; Asthma; Hypersensitivity | interventions — Injections, Subcutaneous; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No immunotherapy, receive standard of care asthma treatment (Active Comparator): This group consists of children who do not receive allergy immunotherapy. Both groups - the experimental as well as the control group receive otherwise standard of care asthma and allergy treatment
  Interventions: Other: Standard of care
- Allergen immunotherapy (Experimental): This group receives initially weekly, later biweekly subcutaneous injections of a mixture of allergen extracts, tailored to the individual child's allergy sensitization profile. The maximum number of injections at each visit is 1-3 injections per child. In addition to allergy immunotherapy. this group receives standard of care asthma and allergy treatment
  Interventions: Biological: Allergen extracts (subcutaneous injections); Other: Standard of care

INTERVENTIONS:
Biological: Allergen extracts (subcutaneous injections) — Allergy immunotherapy consists of regular subcutaneous injections of an individualized mixture of allergen extracts according to the allergy sensitization profile of each child. Increasing doses of allergen extract are given in 1-2 injections until a predetermined maintenance dose is reached. This maintenance dose varies by extract and accords to the general practice guidelines of immunotherapy. To increase safety, the cumulative monthly maintenance doses are divided into biweekly visits during the maintenance phase (year 2-3)
  Arms: Allergen immunotherapy
Other: Standard of care — standard of care asthma and allergy treatment

SUMMARY:
In this clinical study we aim to determine the effect of allergy immunotherapy in decreasing asthma and allergy related disease in children who had multiple episodes of wheezing and who are at high risk for developing persisting asthma. These risks include a history of asthma in the parents, allergies to environmental allergens (such as dust mite, cockroach or mouse) and other allergic diseases such as eczema or food allergies. Allergy Immunotherapy is not new and has been practiced for many years to treat asthma and environmental allergies in older children and adults, but has not yet been systematically studied in young children.

ELIGIBILITY:
Inclusion Criteria:

* Children between 18 months through 3 years who had at least 2 episodes of wheezing prior to enrolment.
* Positive skin tests or specific Immunoglobulin E (IgE) antibody titers to at least one of common airborne allergens: Dust Mite, cat, cockroach, mouse, dog, pollen (all allergy testing can be done at the screening visit at the study site).
* The child must also fulfill the criteria for high risk of developing persistent asthma by meeting at least one of the following major conditions OR 2 of the following minor conditions:

  * Major criteria: History of atopic dermatitis and/or parental history of asthma.
  * Minor criteria: MD-diagnosed allergic rhinitis, wheezing unrelated to colds, blood eosinophils above 4%.

Exclusion Criteria:

* The child has a severe systemic condition (other than allergy or asthma) including (but not limited to) seizures, major congenital anomalies, physical and intellectual delay, cerebral palsy, chest surgery, tuberculosis, primary or secondary immunodeficiency or cardiac disorder (except a hemodynamically insignificant atrial or ventricular septum defect or heart murmur).
* The child was born following 35 or less weeks of gestation.
* Parental report that the child received oxygen for more than 5 days in the neonatal period, or required mechanical ventilation at any time since birth.
* The child fails to thrive, defined as crossing of two major growth percentile lines during the last year.
* The child has chronic lung disease of prematurity (CLDP), cystic fibrosis or any other chronic lung disease.
* The child ever received immunotherapy.
* The child ever received i.v. gammaglobulins or immunosuppressants (other than corticosteroids for asthma).
* History of a life-threatening asthma exacerbation which required intubation and mechanical ventilation.

Ages: 18 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele de Vos, M.D., M.Sc., Principal Investigator — Einstein, Jacobi Medical Center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Abramson MJ, Puy RM, Weiner JM. Allergen immunotherapy for asthma. Cochrane Database Syst Rev. 2003;(4):CD001186. doi: 10.1002/14651858.CD001186. PMID 14583928
- [Background] Roberts G, Hurley C, Turcanu V, Lack G. Grass pollen immunotherapy as an effective therapy for childhood seasonal allergic asthma. J Allergy Clin Immunol. 2006 Feb;117(2):263-8. doi: 10.1016/j.jaci.2005.09.054. PMID 16461125
- [Background] Pifferi M, Baldini G, Marrazzini G, Baldini M, Ragazzo V, Pietrobelli A, Boner AL. Benefits of immunotherapy with a standardized Dermatophagoides pteronyssinus extract in asthmatic children: a three-year prospective study. Allergy. 2002 Sep;57(9):785-90. doi: 10.1034/j.1398-9995.2002.23498.x. PMID 12169173
- [Derived] de Vos G, Viswanathan S, Pichardo Y, Nazari R, Jorge Y, Ren Z, Serebrisky D, Rosenstreich D, Wiznia A. A randomized trial of subcutaneous allergy immunotherapy in inner-city children with asthma less than 4 years of age. Ann Allergy Asthma Immunol. 2021 Apr;126(4):367-377.e5. doi: 10.1016/j.anai.2020.12.016. Epub 2021 Jan 6. PMID 33418053
- [Derived] de Vos G, Nazari R, Ferastraoaru D, Parikh P, Geliebter R, Pichardo Y, Wiznia A, Rosenstreich D. Discordance between aeroallergen specific serum IgE and skin testing in children younger than 4 years. Ann Allergy Asthma Immunol. 2013 Jun;110(6):438-43. doi: 10.1016/j.anai.2013.03.006. Epub 2013 Apr 11. PMID 23706713
- [Derived] de Vos G, Shankar V, Nazari R, Kooragayalu S, Smith M, Wiznia A, Rosenstreich D. Fear of repeated injections in children younger than 4 years receiving subcutaneous allergy immunotherapy. Ann Allergy Asthma Immunol. 2012 Dec;109(6):465-9. doi: 10.1016/j.anai.2012.10.003. PMID 23176889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 children were recruited from one tertiary treatment center, Jacobi Medical Center, which is the largest city hospital in the Bronx, New York. The referral population consists of primarily low-income, Medicaid beneficiaries residing in the Bronx.
Pre-assignment Details: There was no run-in phase. After consents were signed (by the parents), the 58 participants were immediately randomized into treatment or control group. 8 of the 58 participants were withdrawn from the study immediately after randomization, so only 50 participants began protocol treatment.
Groups:
- No Immunotherapy, Receive Standard of Care Asthma Treatment: This group consists of children who do not receive allergy immunotherapy. No placebo injections were used. The control group received standard of care asthma and allergy treatment, excluding allergy immunotherapy (subcutaneous or other routes).
  Standard of care: standard of care asthma and allergy treatment (medications, advice to environmental remediation)
- Allergen Immunotherapy: This group receives initially weekly, later biweekly subcutaneous injections of a mixture of allergen extracts, tailored to the individual child's allergy sensitization profile. The maximum number of injections at each visit is 1-3 injections per child. In addition to allergy immunotherapy, this group receives standard of care asthma and allergy treatment (medications, advice to environmental remediation)
  Allergy immunotherapy consists of regular subcutaneous injections of an individualized mixture of allergen extracts according to the allergy sensitization profile of each child. Increasing doses of allergen extract are given in 1-3 injections until a predetermined maintenance dose is reached. This maintenance dose varies by extract and accords to the general practice guidelines of immunotherapy. To increase safety, the cumulative monthly maintenance doses are divided into biweekly visits during the maintenance phase.
  Standard of care: standard of care asthma and allergy treat
Period: Overall Study
Arm/Group | No Immunotherapy, Receive Standard of Care Asthma Treatment | Allergen Immunotherapy
Started | 27 (4 of 27 withdrew consent immediately after randomization and are excluded from outcome analysis) | 31 (4 of 31 withdrew consent immediately after randomization and are excluded from outcome analysis)
Started Study Protocol (Only participants who started the study protocol were included in the analysis (total n=50)) | 23 | 27
Completed | 17 | 13
Not Completed | 10 | 18
Not completed — Lack of Efficacy | 3 | 6
Not completed — Withdrawal by Subject | 7 | 12

BASELINE CHARACTERISTICS:
Population: Note that of all participants who withdrew from the study, 4 participants in each group (total of 8) withdrew their consent before starting any of the treatment protocol. These 8 withdrawn participants were not included in any analysis.
Groups:
- No Immunotherapy, Receive Standard of Care Asthma Treatment: This group only receives standard of care asthma and allergy treatment. This does not receive allergy immunotherapy.
  Both the experimental group and the control group receive otherwise standard of care asthma and allergy treatment.
- Allergen Immunotherapy: This group receives initially weekly, later biweekly subcutaneous injections of a mixture of allergen extracts, tailored to the individual child's allergy sensitization profile. The maximum number of injections at each visit is 1-3 injections per child. In addition to allergy immunotherapy. this group receives standard of care asthma and allergy treatment
  Allergen extracts (subcutaneous injections): Allergy immunotherapy consists of regular subcutaneous injections of an individualized mixture of allergen extracts according to the allergy sensitization profile of each child. Increasing doses of allergen extract are given in 1-3 injections until a predetermined maintenance dose is reached. For safety, the cumulative monthly maintenance doses are divided into biweekly visits during the maintenance phase.
  Both the experimental group and the control group receive otherwise standard of care asthma and allergy treatment.
- Total: Total of all reporting groups
Arm/Group | No Immunotherapy, Receive Standard of Care Asthma Treatment | Allergen Immunotherapy | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (0.8) | 3.0 (0.8) | 3.1 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 18 | 24 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic/Latino | 15 | 20 | 35
  Ethnicity: Black/African American | 5 | 7 | 12
  Ethnicity: Unknown/not reported | 3 | 0 | 3
Number of children with asthma related Emergency Department visits prior to enrollment [Count of Participants; unit: Participants] | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Asthma Severity as Measured by the Asthma Severity Score (Averaged up to 36 Months)
Description: The Asthma Severity Score is a customized score created for this study due to the lack of standardized instruments for this age group. It takes into account asthma symptom severity and frequency, as well as asthma medication dosing and potency. Data was collected at baseline and every 2 weeks through interviews conducted over the phone. If the caregiver could not be reached by the phone, the interview was conducted at the next face-to face opportunity (study or injection visit). The minimum score on this scale is 0 (no asthma symptoms and no asthma medicines used during the 14 day interview period). The maximum score is 224 (uncontrolled severe asthma with severe cough, shortness of breath and wheezing on 14 of 14 days, using Albuterol 2 puffs 4x/day, budesonide/formoterol 160ug/4.5ug 2 puffs twice daily and Montelukast 4mg daily on 14 of 14 days). Scores calculated from the collected data were averaged to produce one reported value at baseline and year 1, 2 and 3.
Time Frame: baseline and every two weeks up to end of study (up to 36 months)
Population: All participants were included in this analysis that started immunotherapy, regardless if they completed it or not (intention to treat analysis)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | No Immunotherapy, Receive Standard of Care Asthma Treatment | Allergen Immunotherapy
Number analyzed (Participants) | 23 | 27
score on a scale
  Score at baseline | 21.95 (3.74) | 25.68 (3.53)
  Score at Year 1 | 27.72 (3.52) | 27.85 (3.34)
  Score at Year 2 | 31.40 (4.16) | 29.68 (4.03)
  Score at Year 3 | 33.00 (5.23) | 31.15 (5.11)
Statistical Analysis 1: Comparison: Allergen Immunotherapy; Linear mixed effects model (LME) with random coefficients model was fitted with Restricted Maximum Likelihood estimation. The functional form of the model was quadratic and the model adjusted for gender, race, ethnicity and number of asthma hospitalizations since birth. Unequal data collection were smoothed over two month period with a median score values; Test type: Other; p = 0.38, Mixed Models Analysis; Slope = 0.19, 95% CI 2-sided [-0.24 to 0.63], Standard Error of Mean 0.22 — The above is the slope for immunotherapy group . The (quadratic) slope is for 1 month increase in time
Statistical Analysis 2: Comparison: No Immunotherapy, Receive Standard of Care Asthma Treatment; Linear mixed effects model (LME) with random coefficients model was fitted with Restricted Maximum Likelihood estimation. The functional form of the model was quadratic and the model adjusted for gender, race, ethnicity and number of asthma hospitalizations since birth. Unequal data collection were smoothed over two month period with median score values; Test type: Other; p = 0.013, Mixed Models Analysis; The above (quadratic) slope is for control group; Slope = 0.55, 95% CI 2-sided [0.11 to 0.99], Standard Error of Mean 0.22 — The above is the (quadratic) slope is for control group and is for 1 month increase in time
Statistical Analysis 3: Comparison: No Immunotherapy, Receive Standard of Care Asthma Treatment vs Allergen Immunotherapy; Linear mixed effects model (LME) with random coefficients model was fitted with Restricted Maximum Likelihood estimation. The functional form of the model was quadratic and the model adjusted for gender, race, ethnicity and number of asthma hospitalizations since birth. Unequal data collection between immunotherapy and control groups were smoothed over two month period with a median score values; Test type: Other; p = 0.978, contrast testing post mixed model — Post estimation means were tested between the intervention arms after LME model at year 1 and the p- values were adjusted using Bonferroni correction; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-11.76 to 12.03], Standard Error of Mean 4.97 — The difference is IT-Control group and the confidence interval is Bonferroni CI
Statistical Analysis 4: Comparison: No Immunotherapy, Receive Standard of Care Asthma Treatment vs Allergen Immunotherapy; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.77, contrast testing post mixed model] — Post estimation means were tested between the intervention arms after LME model at year 2 and the p- value was unadjusted p value; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-15.83 to 12.38], Standard Error of Mean 5.89 — The difference is IT-Control group and the confidence interval is Bonferroni CI
Statistical Analysis 5: Comparison: No Immunotherapy, Receive Standard of Care Asthma Treatment vs Allergen Immunotherapy; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.80, contrast testing post mixed model — Post estimation means were tested between the intervention arms after LME model at year 3 and the p- values were adjusted using Bonferroni correction; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-19.54 to 15.84], Standard Error of Mean 7.39 — The difference is IT-Control group and the confidence interval is Bonferroni CI

2. Secondary Outcome: Number of Newly Gained Allergic Sensitizations as Assessed by Serum Specific Immunoglobulin E (IgE) Testing
Description: Young children with allergies tend to develop additional environmental allergies over time. This study investigated if allergy immunotherapy could be used to prevent the development of new allergic sensitizations. Participants were tested for sensitivity to a panel of 8 common environmental allergens. Testing was conducted via serum specific immunoglobulin E (IgE) testing. A test was considered negative (non-allergic) if the specific IgE level was <0.35 kIU/L (Kilo International Units/Liter) and positive (allergic) if the levels was >0.35 kIU/L. A "test pair" is the result of a serum IgE test, for a specific allergen, done at two different times. Test pairs can be negative-negative, negative-positive (newly gained allergic sensitization), positive-negative (lost sensitization) or positive-positive. Reported values indicate the total number of newly gained allergic sensitization (negative-positive) for the group.
Time Frame: Baseline and end of treatment (36 months)
Population: In the intention to treat analysis, only 30 children (15 in each group) had serum tests available at baseline and after 36 months of the study.
Measure: Number; unit: Newly gained allergic sensitizations
Units Other Than Participants: test pairs (baseline and at 36+/-6months
Arm/Group | No Immunotherapy, Receive Standard of Care Asthma Treatment | Allergen Immunotherapy
Number analyzed (Participants) | 15 | 15
Number analyzed (test pairs (baseline and at 36+/-6months) | 103 | 105
Newly gained allergic sensitizations | 12 | 16
Statistical Analysis 1: Comparison: No Immunotherapy, Receive Standard of Care Asthma Treatment vs Allergen Immunotherapy; Test type: Superiority; p = 0.677, Chi-squared — Chi-square test (proportion of new sensitizations versus unchanged or lost sensitizations in each group, intention-to treat analysis)

3. Secondary Outcome: Peripheral Blood T Regulatory Cells as a Percentage of CD4+ (Cluster of Differentiation 4) Cells
Description: T regulatory cells are thought to play a role in mediating the effects of immunotherapy in increasing allergen tolerance and dampen the clinical expression of allergy. However, existing studies have not found clear relationship between numbers of T regulatory cells in blood and effect of immunotherapy. The aim of this analysis was to observe potential changes in T regulatory cell numbers in response to immunotherapy in this age group. Peripheral blood cells were acquired and analyzed for T regulatory (Treg) cell markers. In molecular biology, CD4+ (cluster of differentiation 4), a particular cell marker, is a glycoprotein found on the surface of immune cells such as T helper cells and certain groups of T regulatory cells. Testing was done at baseline and then every 12 months. Reported values represents the percentage of CD4+ that are Treg cells.
Time Frame: Baseline and every 12 months until end of treatment (36 months)
Population: Only 27 participants had yearly data for Treg cells from baseline through 36 months (+/- 6 months). Data for 23 participants were not included in the analysis because either parents declined to have blood drawn or because results were not returned from the outside laboratory (despite many efforts to retrieve these data).
Measure: Least Squares Mean (Standard Error); unit: % of CD4+ cells are Treg cells
Groups:
- Allergen Immunotherapy: This group receives initially weekly, later biweekly subcutaneous injections of a mixture of allergen extracts, tailored to the individual child's allergy sensitization profile. The maximum number of injections at each visit is 1-3 injections per child. In addition to allergy immunotherapy. this group receives standard of care asthma and allergy treatment.
  Allergen extracts (subcutaneous injections): Allergy immunotherapy consists of regular subcutaneous injections of an individualized mixture of allergen extracts according to the allergy sensitization profile of each child. Increasing doses of allergen extract are given in 1-3 injections until a predetermined maintenance dose is reached. For safety, the cumulative monthly maintenance doses are divided into biweekly visits during the maintenance phase.
  Both the experimental group and the control group receive otherwise standard of care asthma and allergy treatment.
Arm/Group | No Immunotherapy, Receive Standard of Care Asthma Treatment | Allergen Immunotherapy
Number analyzed (Participants) | 13 | 14
% of CD4+ cells are Treg cells
  Baseline average Treg % | 4.87 (0.65) | 5.90 (0.62)
  1st Year Treg percentage: number analyzed (Participants) | 12 | 10
  1st Year Treg percentage | 5.09 (0.66) | 5.30 (0.73)
  2nd Year Treg percentage: number analyzed (Participants) | 12 | 11
  2nd Year Treg percentage | 5.26 (0.72) | 5.76 (0.74)
  3rd Year Treg percentage | 5.499 (0.92) | 7.08 (0.77)
Statistical Analysis 1: Comparison: No Immunotherapy, Receive Standard of Care Asthma Treatment vs Allergen Immunotherapy; Covariance Pattern Model with autoregressive covariance structure with REML (Restricted Estimation of Maximum Likelihood) with time and role as categorical variable was modeled; Test type: Superiority; p = 0.5460, covariance pattern (rep. measure) model — Test of parallelism (group x time) hypothesis P-value; Within group difference p-values ( baseline vs 3-years) in control and intervention arm were 0.56 and 0.20 respectively; Slope = 0.56, 95% CI 2-sided [-2.18 to 3.29] — The estimated slope reported is for year 3 from the covariance pattern model with autoregressive covariance structure

4. Secondary Outcome: Incidence Rate of Systemic Corticosteroid Bursts (CSB) Per Child
Description: Any reported use of consequent systemic corticosteroid use due to asthma exacerbation counted as one "corticosteroid burst" (CSB). For example, if a child used 5 days of prednisolone due to asthma exacerbation, this counted as one corticosteroid burst (CSB). An interval of at least 7 days was determined to be necessary to count 2 courses of systemic corticosteroids as separated bursts.
  The presented data reflect the intention-to-treat analysis. The time between baseline and each participant's study end time was counted towards the "years in study". The incidence rate describes the number of CSB per child per "year in study".
Time Frame: From baseline through end of study (maximum 36 months)
Population: Participants with available data (intention to treat population)
Measure: Mean (95% Confidence Interval); unit: Number of CSB per child per year
Arm/Group | No Immunotherapy, Receive Standard of Care Asthma Treatment | Allergen Immunotherapy
Number analyzed (Participants) | 23 | 27
Number of CSB per child per year | 1.28 [1.03 to 1.60] | 1.55 [1.26 to 1.90]
Statistical Analysis 1: Comparison: No Immunotherapy, Receive Standard of Care Asthma Treatment vs Allergen Immunotherapy; Null hypothesis = Incidence rate of CSB in each group are same. Poisson regression adjusting for gender, race and history of hospitalization was used to analyze the corticosteroid burst; Test type: Superiority; p = 0.289, Poisson regression — Poisson regression model for treatment arm adjusting for gender, race and history of hospitalization was used to analyze the corticosteroid burst and the time period contributed by each child in years were fitted as offset; Poisson regression model with robust variance with contributed person years used as offset was modeled; Rate ratio = 1.27, 95% CI 2-sided [0.82 to 1.96]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the 3-year study period.
Description: Definition: Serious adverse events= hospitalization, death
  In the immunotherapy group, all allergic or asthmatic events occurring the 48 hours after immunotherapy injections had been administered were considered a possible consequence of immunotherapy (immediate or late allergic reaction). Immediate type reactions were defined as any allergic reaction occurring within 2 hours after the injections.
Groups:
- Allergen Immunotherapy: This group receives initially weekly, later biweekly subcutaneous injections of a mixture of allergen extracts, tailored to the individual child's allergy sensitization profile. The maximum number of injections at each visit is 1-3 injections per child. In addition to allergy immunotherapy. this group receives standard of care asthma and allergy treatment
  Allergen extracts (subcutaneous injections): Allergy immunotherapy consists of regular subcutaneous injections of an individualized mixture of allergen extracts according to the allergy sensitization profile of each child. Increasing doses of allergen extract are given in 1-3 injections until a predetermined maintenance dose is reached. This maintenance dose varies by extract and accords to the general practice guidelines of immunotherapy. To increase safety the cumulative monthly maintenance doses are divided into biweekly visits during the maintenance phase.
  Standard of care: standard of care asthma and allergy treat
Arm/Group | No Immunotherapy, Receive Standard of Care Asthma Treatment | Allergen Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/27
Serious Adverse Events (participants affected / at risk) | 7/23 | 6/27
Other Adverse Events (participants affected / at risk) | 0/23 | 22/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Immunotherapy, Receive Standard of Care Asthma Treatment (N=23) | Allergen Immunotherapy (N=27)
Asthma related hospitalization (Respiratory, thoracic and mediastinal disorders) | 7 (14) | 6 (11) — asthma exacerbation requiring hospitalization
Cellulitis/skin abscess/infected insect bite (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Immunotherapy, Receive Standard of Care Asthma Treatment (N=23) | Allergen Immunotherapy (N=27)
Local allergic reaction after immunotherapy injectionss (Skin and subcutaneous tissue disorders) | 0 | 22 (128) — 22 of 27 (81%): erythema or induration or edema of ≤ 2.5 cm in diameter) 2 of 27 (7%): erythema or induration or edema of > 2.5 cm in diameter but < 50% surface area of upper arm 9 of 27 (33%): mild delayed local reaction
Systemic allergic reactions after immunotherapy injections (Immune system disorders) | 0 | 12 (63) — Systemic reactions were defined as immediate if occurring within 2 hours after injections and delayed if between 2-48 hours after allergy immunotherapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No